CLINICAL TRIAL: NCT01728363
Title: Pharmacokinetics of Antistaphylococcal Antibiotics in Infants
Brief Title: Pharmacokinetics (PK) of Antistaphylococcal Antibiotics in Infants (NICHD-2012-02-Staph Trio)
Acronym: Staph
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phillip Brian Smith (Other)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00037820
Record Dates: First submitted 2012-11-09; First posted 2012-11-19 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Systemic Infection
Keywords: Staphylococcal
MeSH Terms: conditions — Toxemia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ticarcillin-clavulanate antibiotic (Experimental): Cohort Gestational Age (GA) Postnatal Age (PNA) Dose
  1. <30 weeks <14 days: 75 mg/kg Q12 hrs x 6 doses
  2. <30 weeks ≥14 days-45 days 75 mg/kg Q 8 hours x 6 doses
  3. <30 weeks >45 days-90 days 75 mg/kg Q 6 hours x 6 doses
  Brand name is Timentin. This drug is an antibiotic used to treat a wide variety of bacterial infections. It is a combination of two drugs & both treat bacterial infections. Ticarcillin is a penicillin-type antibiotic that stops bacterial growth & clavulanate potassium is an enzyme inhibitor that helps the ticarcillin work better.
  Interventions: Drug: Antibiotic
- Rifampin generic antibiotic (Experimental): Cohort GA PNA Dose
  1. <32 weeks <14 days 10 mg/kg Q 24 hours x 4 doses
  2. <32 weeks ≥14 days-120 days 15 mg/kg Q 24 hours x 4 doses
  3. ≥32 weeks <14 days 15 mg/kg Q 24 hours x 4 doses
  4. ≥32 weeks ≥14 days-120 days 20 mg/kg Q 24 hours x 4 doses
  The brand name is Rifadin, Rimatane. This drug is an antibiotic and a first line antituberculotic and unlabeled use for infections caused by staphylococcus aureus & staphylococcus epidermis.
  Interventions: Drug: Antibiotic
- Clindamycin Generic Antibiotic (Experimental): Cohort GA PNA Dose
  1. <30 weeks <14 days 10 mg/kg Q 12 hours x 6 doses
  2. <30 weeks ≥14 days-45 days 10 mg/kg Q 8 hours x 6 doses
  3. <30 weeks >45 days-120 days 10 mg/kg Q 6 hours x 6 doses
  The brand name is Cleocin. This drug is an antibiotic used to treat a wide variety of bacterial infections and serious infections.
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — Ticarcillin-clavulanate/Timentin is an antibiotic used to treat a wide variety of bacterial infections. Rifampin/Rifadin/Rimatane is an antibiotic and first line antituberculotic. Clindamycin/Cleocin is an antibiotic used to treat a wide variety of bacterial infections and serious bacterial infections.
  Other Names: Ticarcillin-clavulanate generic; Brand Timentin; Rifampin generic; Brand Rifadin, Rimatane; Clindamycin generic; Brand Cleocin

SUMMARY:
Multiple center, open-label, PK study

DETAILED DESCRIPTION:
Pharmacokinetics of rifampin, ticarcillin-clavulanate, and clindamycin antibiotics in hospitalized infants with suspected systemic infection or receiving one of the study drugs per local standard of care. Number of participants are 16-32 evaluable per each study drug of rifampin, ticarcillin-clavulanate, and clindamycin antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient intravascular access
* Suspected systemic infection or receiving 1 of the study drugs per standard of care
* informed consent from legal guardian

Exclusion Criteria:

* history of allergic reaction to study drugs
* urine output <0.5 mL/hr/kg over the prior 24 hours
* serum creatinine >1.7 mg/dl
* Any condition in investigator judgment precludes participation because it could affect participant safety

Ages: 14 Days to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Area under the curve infinity (AUCinfinity) for rifampin | 72 hours
  Pharmacometric analysis of area under the curve at steady state for cohort 1 participants who were dosed with rifampin 10mg/kg Q 24 hours x 4 doses (GA < 32 weeks, PNA < 14 days)
Cohort 1: Maximum concentration (Cmax) of rifampin | 72 hours
  Pharmacometric analysis of maximum concentration after first dose for cohort 1 participants who were dosed with rifampin 10 mg/kg Q 24 hours x 4 doses (GA < 32 weeks, PNA < 14 days)
Cohort 1: Clearance (CL) of rifampin | 72 hours
  Pharmacometric analysis of the clearance for cohort 1 participants who were dosed with rifampin 10 mg/kg Q 24 hours x 4 doses (GA < 32 weeks, PNA < 14 days)
Cohort 1: Volume of distribution at steady state (Vss) of rifampin | 72 hours
  Pharmacometric analysis of volume of distribution at steady state for cohort 1 participants who were dosed with rifampin 10 mg/kg Q 24 hours x 4 doses (GA < 32 weeks, PNA < 14 days)

SECONDARY OUTCOMES:
Cohort 1: Adverse events for participants receiving rifampin | 7 days after last study dose
  Adverse events experienced by cohort 1 participants receiving rifampin 10 mg/kg Q 24 hours x 4 doses (GA < 32 weeks, PNA > 14 days). An adverse event is any untoward medical occurrence in humans, whether or not considered drug-related, that occurs during the conduct of a clinical trial. Any change in clinical status (routine labs, physical examinations, etc.) that is considered clinically significant
Cohort 1 participants: serious adverse events for participants receiving rifampin | 7 days after last study dose
  Serious adverse events experienced by cohort 1 participants receiving rifampin 10 mg/kg Q 24 hours x 4 doses(GA < 32 weeks, PNA > 14 days)Any event that results in any of the following outcomes: death, life-threatening adverse vent, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, inpatient hospitalization or prolongation of existing hospitalization, or important medical event that may jeopardize the health of the study participant or require medical or surgical intervention to prevent another outcome listed above

CONTACTS AND LOCATIONS:
Overall Officials: Philip B Smith, MD, Principal Investigator — Duke Clinical Research Institute and DUMC
Locations (10):
- United States (10):
  - University of FL, Gainesville, Florida
  - UFL Health and Baptist, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wesley Medical, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Kings County Hospital Center, Brooklyn, New York
  - Duke University, Durham, North Carolina
  - University of Texas Children's Hospital, Galveston, Texas

REFERENCES:
- [Background] Maharaj AR, Gonzalez D, Cohen-Wolkowiez M, Hornik CP, Edginton AN. Improving Pediatric Protein Binding Estimates: An Evaluation of alpha1-Acid Glycoprotein Maturation in Healthy and Infected Subjects. Clin Pharmacokinet. 2018 May;57(5):577-589. doi: 10.1007/s40262-017-0576-7. PMID 28779462
- [Result] Gonzalez D, Delmore P, Bloom BT, Cotten CM, Poindexter BB, McGowan E, Shattuck K, Bradford KK, Smith PB, Cohen-Wolkowiez M, Morris M, Yin W, Benjamin DK Jr, Laughon MM. Clindamycin Pharmacokinetics and Safety in Preterm and Term Infants. Antimicrob Agents Chemother. 2016 Apr 22;60(5):2888-94. doi: 10.1128/AAC.03086-15. Print 2016 May. PMID 26926644
- [Result] Smith PB, Cotten CM, Hudak ML, Sullivan JE, Poindexter BB, Cohen-Wolkowiez M, Boakye-Agyeman F, Lewandowski A, Anand R, Benjamin DK Jr, Laughon MM; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Rifampin Pharmacokinetics and Safety in Preterm and Term Infants. Antimicrob Agents Chemother. 2019 May 24;63(6):e00284-19. doi: 10.1128/AAC.00284-19. Print 2019 Jun. PMID 30910891
- [Result] Watt KM, Hornik CP, Balevic SJ, Mundakel G, Cotten CM, Harper B, Benjamin DK Jr, Anand R, Laughon M, Smith PB, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act - Pediatric Trials Network Steering Committee. Pharmacokinetics of ticarcillin-clavulanate in premature infants. Br J Clin Pharmacol. 2019 May;85(5):1021-1027. doi: 10.1111/bcp.13882. Epub 2019 Mar 6. PMID 30710387
- [Result] Smith MJ, Gonzalez D, Goldman JL, Yogev R, Sullivan JE, Reed MD, Anand R, Martz K, Berezny K, Benjamin DK Jr, Smith PB, Cohen-Wolkowiez M, Watt K; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Pharmacokinetics of Clindamycin in Obese and Nonobese Children. Antimicrob Agents Chemother. 2017 Mar 24;61(4):e02014-16. doi: 10.1128/AAC.02014-16. Print 2017 Apr. PMID 28137820

DOCUMENTS (1):
  • Study Protocol (2014-02-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT01728363/Prot_000.pdf